CLINICAL TRIAL: NCT01651234
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Orally Administered GCC-4401C in Healthy Subjects
Brief Title: A Study to Assess Safety, Tolerability, and Pharmacokinetics of Orally Administered GCC4401C in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCC4401C-101
Record Dates: First submitted 2012-07-17; First posted 2012-07-27 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Healthy Male

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: GCC-4401
- Placebo (Placebo Comparator)
  Interventions: Drug: GCC-4401C

INTERVENTIONS:
Drug: GCC-4401 — * Swedish Orange opaque hard gelatin capsules of size 1 with no markings for oral use
  * single dose
  * dosage
    * Cohort 1: 2.5-mg GCC-4401C
    * Cohort 2: 5.0-mg GCC-4401C
    * Cohort 3: 10-mg GCC-4401C
    * Cohort 4: 20-mg GCC-4401C
    * Cohort 5: 40-mg GCC-4401C
    * Cohort 6: 80-mg GCC-4401C
  Arms: Active
Drug: GCC-4401C — * Capsule, identical in appearance to GCC-4401C, for oral use
  * single dose
  * dosage
    * Cohort 1: 2.5-mg matching placebo
    * Cohort 2: 5.0-mg matching placebo
    * Cohort 3: 10-mg matching placebo
    * Cohort 4: 20-mg matching placebo
    * Cohort 5: 40-mg matching placebo
    * Cohort 6: 80-mg matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and characterize the PK, PD f\profile.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the safety and tolerability following administration of single ascending doses of GCC4401C in healthy male subjects; and the secondary objective of this study is to characterize the single-dose PK profile after oral administration of GCC-4401C, and to determine an appropriate dose range and dosing regimen of oral GCC-4401C for subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and complying with the requirements of the study and have signed the informed consent form (ICF);
2. Normal healthy males between 18 and 55 years of age, inclusive, at the time of consent;
3. A body mass index (BMI) of at least 18.5 kg/m2 but no more than 30 kg/m2 (BMI is defined as the subject's weight in kilograms divided by the square root of the subject's height in meters);
4. In general good health based on screening medical history, physical examination (defined as the absence of any clinically significant abnormalities), vital signs, and clinical laboratory values (hematology, serum chemistry, and urinalysis);
5. Have a normal ECG (defined as Fridericia's correction for QT interval [QTcF] less than or equal to 450 ms) at screening, Day -1 and Day 1, predose (baseline). Repeat ECG measurements will be allowed at the baseline assessment for QTcF values above 450 ms and the average will be used to assess eligibility.
6. Male subjects must use barrier contraception during sexual intercourse, ie, condoms, from the first day of dosing until 3 months after the last dosing with GCC-4401C; and
7. Nonsmokers (defined as not having smoked or used any nicotine containing products for at least 1 month, and having a urine cotinine less than 400 ng/mL).

Exclusion Criteria:

Subjects presenting with any of the following will not be entered into the study:

1. Have clinically significant abnormal history, physical findings, or laboratory values at the prestudy screening assessment that could interfere with the objectives of the study or the safety of the subjects;
2. Have any of the following, which may put them at increased risk with anticoagulant use:

   * family history or personal history of bleeding disorders or diseases/syndromes that can either alter or increase the propensity for bleeding;
   * severe trauma, fracture, major surgery, or biopsy of a parenchymal organ within the past 3 months;
   * endoscopic peptic-ulcer disease within the past 3 years or clinically significant gastrointestinal, genitourinary, or gum bleeding within the past 3 months;
   * a personal history of vascular abnormalities including aneurysms; a personal history of severe hemorrhage, hematemesis, melena, hemoptysis, severe epistaxis, severe thrombocytopenia, intracranial hemorrhage; or rectal bleeding within 3 months prior to screening;
   * any history of thrombotic or hemorrhagic stroke;
   * clinically significant laboratory abnormalities (hemoglobin less than 12.0 g/dL, prolonged PT or INR, prolonged aPTT, elevated liver enzymes, elevated serum creatinine or blood urea nitrogen (BUN) which is considered clinically significant by the Investigator, or platelet count less than 150,000/mm3 or greater than 600,000/mm3). Mildly elevated BUN with normal serum creatinine values which are determined not to be clinical significant by the Investigator are permitted. These significant laboratory values may be repeated for confirmation; or
   * any other contraindication to anticoagulant treatment, or increased bleeding risk, as judged by the Investigator.
3. Have known positive test for hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus (HIV) 1, or HIV 2;
4. Are considering or scheduled to undergo any surgical procedure during the study;
5. Have received an investigational product within 30 days prior to dosing;
6. Presence or history of severe adverse reaction to any drug;
7. Involvement in the planning and/or conduct of the study;
8. Positive urine drug screen or urine alcohol screen at medical screening or check-in;
9. History of alcohol, drug, or substance abuse, as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition in the past 12 months;
10. Positive test result for fecal occult blood, measured at screening and/or at check-in to the clinic;
11. Consumption of alcohol within 48 hours prior to dosing;
12. Intake of more than 14 units (a unit is 12 oz beer, 5 oz wine, or 1.5 oz liquor) of alcohol per week;
13. Use of any drugs that induce or inhibit cytochrome P450 or P-glycoprotein within 30 days prior to dosing;
14. Use of any prescribed or over-the-counter (OTC) medications including antacids, analgesics, herbal remedies, vitamins, and minerals (with the exception of up to 3 grams of acetaminophen) or medications containing aspirin or nonsteroidal anti-inflammatory medications with anticoagulant effects within 2 weeks prior to dosing;
15. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of dosing;
16. Planning to father a child or donate sperm during the study and 3 months following dosing;
17. Do not have veins suitable for cannulation or multiple venipunctures;
18. Have previously participated in this study;
19. Donation of plasma or blood products within 1 month of screening or any blood donation/blood loss greater than 450 mL during the 3 months prior to screening; or
20. Any other factor that the Investigator thinks will increase subject risk with participation.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The number and percentage of subjects experiencing 1 or more AEs will be summarized by treatment/dose group, relationship to study drug, and severity. | up to 7 ~ 10 days after administraion
Statistics for clinical laboratory data(continuous variables only), vital signs, and ECF intervals will be presented for each evaluation during the study and for change from baseline to postdose evaluations. | up to 7 ~10 days after administration

SECONDARY OUTCOMES:
the single-dose pharmacokinetic behavior | at predose and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, and 48 hours postdose
  to characterize the single-dose pharmacokinetic behavior after oral administration of GCC-4401C
  * maximum plasma concentration (Cmax);
  * time to Cmax (tmax);
  * terminal rate constant (λz);
  * area under the curve from zero to the time of the last measurable concentration [AUC(0-last)];
  * area under the curve from zero to infinity [AUC(0-inf)];
  * apparent terminal half-life (t½);
  * apparent systemic clearance (CL/F);
  * apparent volume of distribution (Vz/F);
  * renal clearance (CLr); and
  * fraction of drug (fe) excreted unchanged in urine (% of dose).

OTHER OUTCOMES:
the single-dose pharmacodynamics behavior | at predose and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, and 48 hours postdose
  * PT;
  * aPTT;
  * INR;
  * coagulation factor X assay;
  * If the assay for coagulation factor X is abnormal a reflex inhibitor screen will be performed. This test will not be run on coagulation factor X assay results which are within normal range.
  * anti factor Xa assay;
  * escarin-stimulated thrombin activity; and
  * antithrombin (III) activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phase1 Unit, Overland Park, Kansas, United States